CLINICAL TRIAL: NCT01848964
Title: Peut-on améliorer la Marche de l'amputé fémoral en Guidant la Correction prothétique Par l'Analyse Des Pressions Dans l'emboîture ?
Brief Title: Analyzing Stump-socket Interface Pressure to Improve Gait in Above-knee Amputee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A00219-36
Record Dates: First submitted 2013-04-19; First posted 2013-05-08 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: amputation; prosthesis; stump; socket; pressure; gait; posture
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Evaluation (Experimental): First, the assessment will be performed to evaluate the relationship between pressure repartition pattern, clinical evaluation and motor capabilities. All the patients and volunteers will be concerned by this first part.
  A second part will be conducted in 15 amputees within the 40 patients. Assessments of pressure pattern during gait and standing will be repeated two times: by the same investigator and by a different investigator, in order to test intra- and inter-evaluator reproducibility.
  After the first assessment, the prosthesis may be modified in order to solve clinical problems. In that case, a new assessment will be proposed 2 to 8 weeks after in order to test the effect of the prosthesis modification on pressure pattern, gait, posture and clinical parameters.
  Interventions: Device: Clinical and instrumented measurements

INTERVENTIONS:
Device: Clinical and instrumented measurements — Clinical examination will include stump pain, wound, scar and unusual shape.
  Questionnaire will include satisfaction scale (SatPro), comfort scale (SCE), and functional scale (PPA-LCI)
  After installing the sensors on the stump, the patient will put his prosthesis on and will perform the following tasks: gait, sitting and standing posture and gait initiation.
  Pressure repartition at the stump-socket interface will be assessed with the 14 flat sensors.
  Gait parameters will be assessed with the OptoGait device. Standing posture and gait initiation parameters will be assessed with a force-plate.

SUMMARY:
This study aims at evaluating the relation between quality of the interface between the stump and the prosthesis, and the quality of gait in above-knee amputees.

The hypothesis is that an adapted prosthesis allowing an efficient gait in above-knee amputees corresponds to an homogeneous pressure distribution pattern onto the stump.

DETAILED DESCRIPTION:
Forty amputee patients will be evaluated for satisfaction with the prosthesis, pressure repartition pattern and functional capabilities.

Pressure at the stump-socket interface will be recorded using a set of 14 single cells sensors placed in predefined positions onto the stump. Pattern of pressure will be measured in four tasks: sitting posture, standing posture, gait initiation, and gait at preferred velocity.

Reproducibility of the pressure repartition pattern will be analyzed by repeating gait and standing posture task in the first 15 patients included.

In patients whom prosthesis has been modified on the basis on the first pressure measurement (pressure peak and bad functional capacities), a new pressure measurement will be repeated 2-8 weeks apart.

Postural and gait abilities will be also assessed in 40 age/gender matched non-amputated subjects to serve as control data.

ELIGIBILITY:
1. Amputee patients:

   Inclusion Criteria:
   * unilateral transfemoral amputation
   * use of a prosthesis with a "contact" socket

   Exclusion Criteria:
   * neurological or muscular disorder likely to impair walking capabilities
   * Mini Mental State Examination below 24/30
2. Healthy subjects :

Exclusion Criteria:

* neurological or muscular disorder likely to impair walking capabilities
* Mini Mental State Examination below 24/30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Two minute Walking Test | At inclusion (baseline) for all patients
  Maximal distance(m)walked during 2 minutes (one trial)

SECONDARY OUTCOMES:
Variation coefficient of maximal pressures during gait | At inclusion (Baseline) for all patients
  Calculated on the basis of 10 walking trials of 10 meters. The maximal pressure will be measured at each step for each sensor. The mean maximal pressure is calculated for each of the 14 sensors. The variation coefficient is calculated between these 14 values (variation coefficient = standard deviation/mean)
  A low variation coefficient of pressure is supposed to represent an homogeneous repartition of the pressure in the prosthesis.
Change in two minutes walk tests between Baseline and 5 Weeks | Five weeks (W5) in average after inclusion in patients in whom the prosthesis will be modified
  If a modification of the prosthesis is required and performed on the basis of the first assessment (at inclusion), a new assessment with the modified prosthesis is performed 5 weeks later (from 2 to 8 weeks).
  Change in walking capabilities is assessed by calculating the difference between results of the two minute walk test at inclusion and at 5 weeks.
Change in the variation coefficients of maximal pressures between Baseline and 5 Weeks | 5 Weeks in average (2 and 8 weeks) after the inclusion in patients in whom the prosthesis will be modified
  If a modification of the prosthesis is required and performed on the basis of the first assessment (at inclusion), a new assessment with the modified prosthesis is performed 5 weeks later (from 2 to 8 weeks).
  Change of repartition pattern will be assessed by calculating the difference between the variation coefficient before and after the prosthesis modification.
Gait spatial and temporal parameters | At inclusion for all patients
  Calculated based on 10 walking trial of 10 meters. Speed, step length of the prosthetic and non-amputated leg and standing time on the prosthetic and non-amputated leg
Variation coefficient of maximal pressure during standing posture | At inclusion for all patients
  Calculated based on 4 standing trial of 30 seconds. The calculation is the same as for gait, but the mean pressure during the postural trial will be used instead of the maximal pressure during the step.
Reproducibility of the Variation Coefficients of maximal pressures | At baseline
  At inclusion (baseline), the measurements of pressure repartition pattern in gait and standing posture tasks will be repeated twice, in order to test inter- and intra-evaluator reproducibility.

OTHER OUTCOMES:
Occurrence of pain, dyscomfort, or skin wound due to the measurement system | at baseline
  By structured interview, visual analogic pain scale, and clinical examination at the end of the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Pérennou, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France